CLINICAL TRIAL: NCT02260336
Title: The Effect of Panax Notoginseng Powders on Rheumatic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chengdu PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yang Min, Ph.D, Chengdu PLA General Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PNP01RP001
Record Dates: First submitted 2014-10-03; First posted 2014-10-09 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Rheumatic Pain
MeSH Terms: conditions — Musculoskeletal Pain | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Panax Notoginseng Powder 1g (Experimental): Panax Notoginseng Powder 1g, daily
  Interventions: Dietary Supplement: Panax Notoginseng Powder 1g
- Panax Notoginseng Powder 5g (Experimental): Panax Notoginseng Powder 5g,daily
  Interventions: Dietary Supplement: Panax Notoginseng Powder 5g
- Panax Notoginseng Powder 10g (Experimental): Panax Notoginseng Powder 10g,daily
  Interventions: Dietary Supplement: Panax Notoginseng Powder 10g
- Panax Notoginseng Powder 15g (Experimental): Panax Notoginseng Powder 15g,daily
  Interventions: Dietary Supplement: Panax Notoginseng Powder 15g
- Celecoxib Capsule 400 mg daily (Active Comparator): Celecoxib Capsule 400 mg daily
  Interventions: Drug: Celecoxib Capsule 400 mg daily

INTERVENTIONS:
Dietary Supplement: Panax Notoginseng Powder 1g
  Arms: Panax Notoginseng Powder 1g
Dietary Supplement: Panax Notoginseng Powder 5g
  Arms: Panax Notoginseng Powder 5g
Dietary Supplement: Panax Notoginseng Powder 10g
  Arms: Panax Notoginseng Powder 10g
Dietary Supplement: Panax Notoginseng Powder 15g
  Arms: Panax Notoginseng Powder 15g
Drug: Celecoxib Capsule 400 mg daily
  Arms: Celecoxib Capsule 400 mg daily

SUMMARY:
The purpose of this study is to evaluate the effect of Panax Notoginseng Powders on Rheumatic Pain.

ELIGIBILITY:
Inclusion Criteria:

* had a diagnosis of classic or definite RA
* without conflict to the written, informed consent signed prior to the enrollment.

Exclusion Criteria:

* uncontrolled medical problems
* organic brain syndrome
* major psychiatric disturbances
* major communicative disorders
* a history of severe noncompliance
* less than 7 years of formal education, or illiteracy
* being included in other clinical trial within the last 4 weeks
* with abnormal liver or kidney function (more than 1 time above the high normal)
* with serious cardiovascular disease
* with hematologic disease
* being in pregnancy, lactation period or under a pregnancy plan
* with severe gastrointestinal disease
* with contraindication or being allergic to the test drugs
* being under the treatment of drugs within 1 previous week, that might affect the results of the trial, such as non-steroidal anti-inflammatory drugs
* being not compatible for the trial medication, or other circumstances at the discretion of investigators
* without legal capacity or only with limited legal capacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in McGill Pain Questionnaire (MPQ) score at 24 weeks | at 0 week, 6 weeks, 12 weeks, 24 weeks
  This well validated questionnaire assesses pain on several dimensions including sensory pain, affective pain, and evaluative pain.
Change from Baseline in Visual Analog Scale(VAS) score at 24 weeks | at 0 week, 6 weeks, 12 weeks, 24 weeks
  This rating scale involved the selection of a point along a 10-cm line, which described pain intensity on a continuum from "no pain at all" to "pain as bad as it could be." This scale has been found to be an excellent measure of self-reported pain

CONTACTS AND LOCATIONS:
Locations (1):
- 270 Rongdu street, Jin-niu district,Rheumatology Center of Integrated Medicine, General Hospital of Chengdu Military Area Command PLA，, Chengdu, Sichuan, China